CLINICAL TRIAL: NCT01225783
Title: The Validity and Reliability of Self Measurement of Upper Limb Volume in Treating Lymphedema in Breast Cancer Patients
Brief Title: The Validity and Reliability of Self Measurement of Upper Limb Volume
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMC10095KCTIL
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Limb Volume Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Self measurement of limb volume +water displacement — Comparison will be made between self measurement is two types of tape measure compared with water displacement

SUMMARY:
Lymphedema is a common, chronic, side effect resulting from the treatment of breast cancer.Insufficiency in the lymphatic system causes edema in the upper limb. The accepted conservative treatment is based on the anatomy and physiology of the lymphatic system. The aim of the treatment is to reduce the volume of the upper limb by, initial, intensive treatment and then to keep the arm volume at this reduced level.The measurement of limb volume involves measuring the circumference of the arm at defined points and then with the use of a formula the volume of the arm can be calculated. After intensive therapy is complete the responsibility for measuring limb volume moves to the patient. This study will examine the reliability and validity of self measurement of limb volume. The investigators will compare the results of self measurement using the accepted plastic tapemeasure against a paper tape measure adapted for self measurement.Both methods will be compared to the "gold standard volume displacement. In the study there will be two meetings with the subjects where the patient and physiotherapist will use the three methods.

ELIGIBILITY:
Inclusion Criteria:

* Women with arm edema after breast cancer who are being conservatively treated by a physiotherapist.

Exclusion Criteria:

* Active malignant disease

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of self measurement of limb volume to water displacement | 2 years
validity of self measurement | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Remez Health center, Rehovot, Israel